CLINICAL TRIAL: NCT01995227
Title: An Individualized Anti-Cancer Vaccine (AlloVaxTM) Study in Patients With Refractory Hepatocellular Carcinoma (HCC)
Brief Title: An Individualized Anti-Cancer Vaccine Study in Patients With HCC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study site change to Thailand
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-019-HCC-VAX
Record Dates: First submitted 2013-11-18; First posted 2013-11-26 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2015-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; HCC; tumor vaccine; immunotherapy; personalized anti-cancer vaccine
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AlloVax Treatment (Experimental): Intradermal injection (ID) of AlloStim(TM) (1ml) on day 4 and 7. AlloVax Treatment: ID injection of AlloSim(TM) (1 ml) followed immediately by the ID injection of CRCL (1ml) on day 11 and 14 in same location on the left arm and on day 18 and 21 in the same location on the right arm. Intravenous infusion of AlloStim(TM)(5ml) and a CRCL alone Intradermal injection on Day 27.
  Interventions: Biological: AlloVax; Biological: CRCL; Biological: AlloStim

INTERVENTIONS:
Biological: AlloVax — Personalized anti-cancer vaccine
  Other Names: AlloStim plus CRCL
Biological: CRCL — Personalized anti-cancer vaccine
  Other Names: Chaperone Rich Cell Lysate; AlloVax
Biological: AlloStim — ID injections IV infusion
  Other Names: AlloStim ID; AlloStim IV

SUMMARY:
The purpose of this study is to determine the safety and the immunological, radiological, and pathological response of the personalized anti-cancer vaccine AlloVax(TM) in patients with refractory Hepatocellular Carcinoma (HCC) and who are not eligible for any approved HCC treatments or have failed all approved HCC treatments. AlloVax(TM) is a personalized anti-cancer vaccine combining Chaperone Rich Cell Lysate (CRCL) as a source of tumor antigen prepared from patient's tumor and AlloStim(TM) as an adjuvant. The combination of these two components provides a vaccine designed to bring out an immune response capable of finding and killing the tumor cells.

DETAILED DESCRIPTION:
All accrued subjects will undergo tumor harvest procedure. The tumor samples will be processed into personalized Chaperone Rich Cell Lysate (CRCL) vaccine. This study consists of three phases: priming phase, vaccination phase, and activation phase. The priming phase involves intradermal injections of AlloStim(TM). The aim of this phase is to increase the titer of Th1 immune cells in circulation. The vaccination phase involves the intradermal injections of AlloSim(TM) immediately followed by the intradermal injections of CRCL. This phase is designed to elicit tumor-specific immunity. The activation phase involves intravenous infusion of AlloStim(TM). This phase is designed to activate memory cells and NK cells and cause them to extravasate and traffic to tumor sites.

ELIGIBILITY:
Inclusion Criteria:

* Any Patients with a diagnosis of HCC based on histology or the current accepted radiological measures.
* Age > 18 years.
* Patient has an MRI or CT result (positive for HCC) up to 3 months prior to recruitment.
* AFP > 30.
* Patient who is not eligible or failed all approved HCC treatments.

Exclusion Criteria:

* Patient is unable or unwilling to sign informed consent.
* Patients that are participating in other clinical trials evaluating experimental treatments or procedures.
* Severe congestive heart failure (LVEF on echocardiogram < 20%).
* Severe pulmonary hypertension (By echocardiogram, PAS >45 mmHg).
* Uncontrolled diabetes mellitus (HBA1C >9.5%).
* Any autoimmune disorder, which is currently being treated with prednisone or any other immune suppressive medication.
* Patients currently receiving total parenteral nutrition if they have contraindications to oral drugs.
* Patients with positive HIV1, HIV2, HTLV1, HTLV2, and RPR (syphilis).
* Women who are pregnant or breast feeding.
* Patients, based on the opinion of the investigator, should not be enrolled into this study.
* HBV DNA positive.
* If the patient is HBsAg positive or HBcAB positive, but HBV DNA negative, irrespective of his/her anti-HBS status, patient can be enrolled, but will receive preemptive therapy with Lamivudine.
* Patients with HBV DNA positive will not be enroll, but if turned negative with therapy can be enrolled. Patients with HBV and HCV will be followed by HBV DNA and HCV RNA levels during the trial.
* Any metastasis except for portal vein involvement.
* Patients with Child Pugh above B8.
* Prior experimental therapy or cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine).
* History of blood transfusion reactions.
* Known allergy to bovine or murine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2018-02 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Safety | 30 days
  To assess adverse events and laboratory abnormalities associated with AlloVax

SECONDARY OUTCOMES:
Tumor-Specific Immunity | 30 days
  Determine if AlloVax elicits detectable tumor specific immunity
Tumor Biomarker Status | 30 days
  Biomarker concentration will be evaluated at different time points.

OTHER OUTCOMES:
Anti-Tumor Response | 30 days
  To determine if there are any evidence of anti-tumor immune-mediated response by radiological and pathological changes.
Overall Survival (OS) | approximately 12 months
  Baseline to date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hebrew University-Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Result] Epple LM, Bemis LT, Cavanaugh RP, Skope A, Mayer-Sonnenfeld T, Frank C, Olver CS, Lencioni AM, Dusto NL, Tal A, Har-Noy M, Lillehei KO, Katsanis E, Graner MW. Prolonged remission of advanced bronchoalveolar adenocarcinoma in a dog treated with autologous, tumour-derived chaperone-rich cell lysate (CRCL) vaccine. Int J Hyperthermia. 2013 Aug;29(5):390-8. doi: 10.3109/02656736.2013.800997. Epub 2013 Jun 20. PMID 23786302
- [Result] Mayer-Sonnenfeld T, Har-Noy M, Lillehei KO, Graner MW. Proteomic analyses of different human tumour-derived chaperone-rich cell lysate (CRCL) anti-cancer vaccines reveal antigen content and strong similarities amongst the vaccines along with a basis for CRCL's unique structure: CRCL vaccine proteome leads to unique structure. Int J Hyperthermia. 2013 Sep;29(6):520-7. doi: 10.3109/02656736.2013.796529. Epub 2013 Jun 4. PMID 23734882
- [Result] LaCasse CJ, Janikashvili N, Larmonier CB, Alizadeh D, Hanke N, Kartchner J, Situ E, Centuori S, Har-Noy M, Bonnotte B, Katsanis E, Larmonier N. Th-1 lymphocytes induce dendritic cell tumor killing activity by an IFN-gamma-dependent mechanism. J Immunol. 2011 Dec 15;187(12):6310-7. doi: 10.4049/jimmunol.1101812. Epub 2011 Nov 9. PMID 22075702
- [Result] Janikashvili N, LaCasse CJ, Larmonier C, Trad M, Herrell A, Bustamante S, Bonnotte B, Har-Noy M, Larmonier N, Katsanis E. Allogeneic effector/memory Th-1 cells impair FoxP3+ regulatory T lymphocytes and synergize with chaperone-rich cell lysate vaccine to treat leukemia. Blood. 2011 Feb 3;117(5):1555-64. doi: 10.1182/blood-2010-06-288621. Epub 2010 Dec 1. PMID 21123824
- [Result] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Result] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- See also: Liver Cancer — http://www.nlm.nih.gov/medlineplus/livercancer.html